CLINICAL TRIAL: NCT06060366
Title: Impact of Pulmonary Endarterectomy on Sleep-Related Breathing Disorders and Mortality in Chronic Thromboembolic Pulmonary Hypertension - The IPES Trial: A Prospective, Observational, Cohort Study
Brief Title: Impact of Pulmonary Endarterectomy on Sleep-Related Breathing Disorders in CTEPH: The IPES Trial
Acronym: IPES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 20231009
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Sleep-Disordered Breathing; Chronic Thromboembolic Pulmonary Hypertension; Post Operative
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PE for CTEPH: CTEPH patients who were eligible for operation
  Interventions: Procedure: Pulmonary endarterectomy
- Medical treatment CTEPH: CTEPH patients who were not eligible for surgery of any reason and decided to follow up with medical treatment

INTERVENTIONS:
Procedure: Pulmonary endarterectomy — removal of chronic thrombus from pulmonary arterial system
  Groups: PE for CTEPH

SUMMARY:
Pulmonary hypertension (PH) has three main types, pre-capillary PH, post-capillary PH, and combined pre-capillary and post-capillary PH, and it is based on mean pulmonary arterial pressure (PAP) > 20 mmHg measured with a right heart catheterization (RHC).

Chronic thromboembolic pulmonary hypertension (CTEPH) is mainly defined as a pre-capillary PH and classed as a Group IV PH. It was reported that 0.1-9.1% of individuals with pulmonary embolism develop CTEPH within two years after the initial diagnosis, and CTEPH is the only PH category that has a chance of being cured, mainly by pulmonary endarterectomy.

Sleep-related breathing disorders (SRBD) are defined as obstructive sleep apnea (OSA) disorders, central sleep apnea (CSA) syndromes, sleep-related hypoventilation disorders, and sleep-related hypoxemia.

An SRBD may also lead to an increase in PAP primarily during sleep and cause nocturnal hypoxemia. Although SRBDs were reported in patients with pre-capillary PH, most of the studies included patients with idiopathic PAH. Although the cause-and-effect relationship between pre-capillary PH and SRBDs is uncertain, it is known that mPAP may increase during sleep in patients with OSA .

Less is known regarding the occurrence of SRBDs in CTEPH. Previously a few study showed relationship between SRBDs an CTEPH as the main type was OSA. Most of the studies evaluated preoperative occurance and incidance of SRBDs in CTEPH. Only one study performed post operative SRBD on a cardiorespiratory device was conducted the night before and one month after elective pulmonary endarterectomy.

In our previous study we showed that severe nocturnal hypoxemia (NH) is highly prevelant in preoperative CTEPH patients and the most common two types of SRBD are OSA and isolated sleep related hypoxemia (ISRH) and age, mPAP and AHI are independent determinants of severe NH. (J. Clin. Med. 2023, 12, 4639 https://doi.org/10.3390/jcm12144639) In this present study we aimed to investigate occurrence of SRBDs and mortality 5 years after pulmonary endarterectomy operation.

DETAILED DESCRIPTION:
This study planned as continuation study of ''Determinants of severe nocturnal hypoxemia in adults with chronic thromboembolic pulmonary hypertension and sleep related breathing disorders'' J. Clin. Med. 2023, 12, 4639 https://doi.org/10.3390/jcm12144639

Previously included patients (50 patients who were referred for pulmonary endarterectomy operation between 5 May 2017 and 7 February 2018

* All participants underwent a computerized pulmonary angiography and RHC after that mismatch of perfusion defects detected in ventilation/perfusion scintigraphy (V/Q) despite 3 months of anticoagulant therapy.
* Patients with an mPAP > 20 mmHg measured with RHC were accepted having CTEPH PAWP≤15mmHg and PVR≥ 3 Wood Units were additional measurements suggestive of CTEPH.
* Eligible for surgery
* Appropriate polisomnography test before surgery

  * Total sleep time should be >4 hours) planned to include current study

    1. Demographic data, body mass index (BMI), comorbid conditions, medications, supplementary oxygen treatment, preoperative echocardiography findings, RHC measurements, 6 min walk distance (SMWD), pulmonary function test, as well as carbon monoxide diffusion test (DLCO) measurements will be recorded

       **MIR Spirolab II spirometry (Medical International Research, Rome, Italy) was used to test pulmonary function, including forced expiratory volume in one second (FEV1) and forced vital capacity (FVC), diffusing capacity of the lung for DLCO in a body plethsmograph (CareFusion Type MasterScreen PFT, Hoechberg, Germany), and performance of an SMWD. All results were assessed in accordance with ATS recommendations
    2. A polisomnography test will perfomed to all participants (whether had pulmonary endarterectomy operation or followed up by medical treatment)

       * All patients will hospitalized for polysomnographic monitoring using the NOX- A1 system (Nox Medical Inc., Reykjavik, Iceland). The PSG recording included an elec- troencephalogram (F4/M1, F3/M2, C4/M1, C3/M2, O2/M1, O1/M2), electro-oculogram, submental and tibialis electromyograms, as well as an electrocardiogram. Ventilatory monitoring included a nasal pressure detector using a nasal cannula/pressure transducer system and thoracoabdominal movement detection through two respiratory inductance plethysmography belts. A finger pulse oximeter detecting heart rate, SpO2, as well as body position and movement detection will also include. Participants with a total sleep time of less than 4 h will be offered a new PSG. Sleep stages and arousals will score based on 30 s epochs in accordance with The AASM Manual for the Scoring of Sleep and Associated Events 2.5 published by the American Academy of Sleep Medicine (AASM), independently of the patients' clinics, by a certified sleep physician. Apnea will define as an almost complete (≥ 90%) cessation of airflow, and hypopnea will define as a decrease in nasal pressure amplitude of 30% or more and/or thoraco-abdominal movement of at least 30% for at least 10 s if there will be a significant oxyhemoglobin desaturation (reduction of at least 3% from the immediately preceding baseline value) and/or arousal, according to the latest recommendations of the AASM
       * SRBDs defined according to the International Classification of Sleep Disorders (ICSD)-10 as obstructive sleep apnea (OSA; as an AHI ≥ 15 events/h), central sleep apnea with Cheyne-Stokes respiration (CSA-CSR; CSR pattern ≥ 50% of total sleep time with , (TST)), obesity hypoventilation syndrome (OHS), and isolated sleep-related hypoxemia (ISRH) (nocturnal oxyhemoglobin saturation (SpO2) < 88% for 5 min or more without OSA, CSA, or OHS) Severe NH was defined as SpO2 < 90% for more than 20% of total sleep time (TST)
    3. Cardiac evaluation will be performed by transthoracic-echocardiography (TTE) TTE based on the guidelines of the device (Epiq 7, Philips Healthcare, Andover, MA, USA) with a 3.5 MHz (S5-1) transducer. Digitally stored images will analyze offline (Xcelera, Philips). Based on the guidelines, the systolic and diastolic characteristics of the left and right heart will measure as recommended. Tricuspid regurgitation velocity and other echocardiographic signs will combine to assess the probability of PH as recommended in ERS guidelines

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with CTEPH according to radiology and right heart catheterization and eligible for surgery
* Polisomnography test
* Includes both criteria above

Exclusion Criteria:

* do not volunter for study
* exitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be the same in our previous which was mentioned above
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  mortality of patients who were or operated or followed up by medical treatment

SECONDARY OUTCOMES:
Type of Sleep-Related Breathing Disorders | 5 years
  Type of the SRBD after operation ar medical treatment
systolic pulmonary arterial pressure (sPAP) | 5 years
  Change in sPAP by transthoracic echocardiography after surgery or medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sehnaz Olgun Yildizeli, Assoc Prof, Principal Investigator — ICJME
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, Williams PG, Souza R. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801913. doi: 10.1183/13993003.01913-2018. Print 2019 Jan. PMID 30545968
- [Result] Badesch DB, Raskob GE, Elliott CG, Krichman AM, Farber HW, Frost AE, Barst RJ, Benza RL, Liou TG, Turner M, Giles S, Feldkircher K, Miller DP, McGoon MD. Pulmonary arterial hypertension: baseline characteristics from the REVEAL Registry. Chest. 2010 Feb;137(2):376-87. doi: 10.1378/chest.09-1140. Epub 2009 Oct 16. PMID 19837821
- [Result] Madani MM. Pulmonary endarterectomy for chronic thromboembolic pulmonary hypertension: state-of-the-art 2020. Pulm Circ. 2021 May 24;11(2):20458940211007372. doi: 10.1177/20458940211007372. eCollection 2021 Apr-Jun. PMID 34104418
- [Result] La Rovere MT, Fanfulla F, Taurino AE, Bruschi C, Maestri R, Robbi E, Maestroni R, Pronzato C, Pin M, D'Armini AM, Pinna GD. Chronic thromboembolic pulmonary hypertension: Reversal of pulmonary hypertension but not sleep disordered breathing following pulmonary endarterectomy. Int J Cardiol. 2018 Aug 1;264:147-152. doi: 10.1016/j.ijcard.2018.02.112. PMID 29776563
- [Result] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376
- [Result] Cinar C, Yildizeli SO, Balcan B, Yildizeli B, Mutlu B, Peker Y. Determinants of Severe Nocturnal Hypoxemia in Adults with Chronic Thromboembolic Pulmonary Hypertension and Sleep-Related Breathing Disorders. J Clin Med. 2023 Jul 12;12(14):4639. doi: 10.3390/jcm12144639. PMID 37510754